CLINICAL TRIAL: NCT06775899
Title: Evaluating the Efficacy of a Cost-Effective PC-Based Tool as a Non-Inferior Alternative to Traditional Ultrasound Simulators in Medical Education
Brief Title: Equivalence Study Comparing a Cost-Effective PC-Based Ultrasound Training Tool to Traditional Simulators in Third-Year Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Samuel Agostino, PhD, Research Technician, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 219864
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Ultrasound; Medical Training; Simulation Based Learning; Medical Student
Keywords: Medical Education; Ultrasound Simulation; PC-Based Training Tool; Thoracic Ultrasound; Abdominal Ultrasound; Cost-effective Simulator; Clinical Skills Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulator Thoracic and Abdominal (Active Comparator): Participants in this group will receive ultrasound training using a traditional, medium-cost ultrasound simulator (VausSim). This simulator allows students to practice image acquisition and pathology recognition in a controlled environment. Training will also include hands-on practice with healthy volunteers. The performance of students in this group will be compared to those using the PC-based tool to determine if both methods produce similar learning outcomes.
  Interventions: Device: Traditional Ultrasound Simulator (VausSim)
- PC-based tool (Experimental): Participants in this group will receive ultrasound training using an interactive PC-based tool. This tool provides real ultrasound images and videos to simulate pathology recognition and image optimization. Students will rotate through different training stations, including hands-on practice with healthy volunteers. The goal is to assess whether this low-cost digital tool is as effective as a traditional ultrasound simulator for teaching ultrasound skills.
  Interventions: Device: PC-Based Ultrasound Training Tool

INTERVENTIONS:
Device: PC-Based Ultrasound Training Tool — An interactive, PowerPoint-based PC tool designed to simulate pathology recognition and ultrasound image optimization for medical students. It provides real ultrasound videos and images, allowing students to practice diagnostic interpretation and image acquisition in a structured training format.
  Arms: PC-based tool
Device: Traditional Ultrasound Simulator (VausSim) — A medium-cost ultrasound simulator used for hands-on training in thoracic and abdominal ultrasound. It allows medical students to practice probe handling, image acquisition, and pathology recognition in a controlled simulation environment.
  Arms: Simulator Thoracic and Abdominal

SUMMARY:
Brief Summary:

The goal of this clinical trial is to determine if a cost-effective, PC-based ultrasound training tool is as effective as a traditional, medium-cost ultrasound simulator for teaching third-year medical students thoracic and abdominal ultrasound skills. This study focuses on improving access to high-quality ultrasound training in educational settings with limited resources. The main questions it aims to answer are:

1. Does the PC-based tool help participants improve their ability to optimize ultrasound images in a way comparable to the traditional simulator?
2. Can participants using the PC-based tool identify and interpret pathological conditions with the same accuracy as those using the traditional simulator?

Participants are third-year medical students enrolled in a structured internship. They will:

1. Watch educational videos covering key concepts in thoracic and abdominal ultrasound imaging.
2. Rotate through training stations where they will practice using either the PC-based tool or the traditional simulator.
3. Perform hands-on exercises with healthy volunteers to practice image acquisition and recognition of anatomical structures.
4. Complete pre- and post-training assessments to measure their progress in skills such as image optimization and identifying pathological conditions.

This study aims to explore whether a low-cost digital solution can provide equal educational value, offering a practical alternative to traditional simulators in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Third-year medical students enrolled in the "Approach to Ultrasound" internship.
* Participants who have completed the preliminary blended learning videos on thoracic and abdominal ultrasound techniques.
* Participants with or without prior minimal experience in using an ultrasound probe, provided they have not undergone formal specialized ultrasound training.

Exclusion Criteria:

* Inability to attend all training sessions and assessments as per the study schedule.
* Physical or medical conditions that limit the ability to perform hands-on ultrasound practice (e.g., musculoskeletal injuries).
* Refusal to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Improvement in Image Optimization Skills | Measured immediately before and after the training session.
  Change in the Objective Structured Assessment of Ultrasound Skills (OSAUS) scores for image optimization pre- and post-training.
Pathology Recognition Accuracy | Measured immediately before and after the training session.
  Change in the ability to identify and interpret pathological ultrasound images, scored on a scale of 0-3 (0 = no recognition, 3 = full recognition).

SECONDARY OUTCOMES:
Participant Satisfaction with Training | Measured immediately after the training session.
  Participant satisfaction assessed through a Likert-scale questionnaire (1-5, where 5 = very satisfied).
Time Required for Image Acquisition | Measured immediately before and after the training session.
  Change in the time taken to acquire specific ultrasound views in healthy volunteers and pathology recognition (measured in seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- SimTo Advanced Medical Simulation Centre, Turin, Italy, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared at this time because additional analyses and follow-up studies are currently in progress. Future research will further explore the implications of the findings, and data sharing may be reconsidered once all related studies are completed and published

REFERENCES:
- [Background] Kollmann C, Flor M, Bader R. A web-based modern ultrasound diagnostic scanner simulation (SimulUS) for undergraduate medical e-learning education. Med Ultrason. 2016 Sep;18(3):408-9. doi: 10.11152/mu.2013.2066.183.kol. No abstract available. PMID 27622424
- [Background] Weimer J, Recker F, Hasenburg A, Buggenhagen H, Karbach K, Beer L, Weimer A, Schiestl L, Lorenz L, Kloeckner R, Dionysopoulou A. Development and evaluation of a "simulator-based" ultrasound training program for university teaching in obstetrics and gynecology-the prospective GynSim study. Front Med (Lausanne). 2024 Apr 24;11:1371141. doi: 10.3389/fmed.2024.1371141. eCollection 2024. PMID 38721350
- [Background] Pezel T, Dreyfus J, Mouhat B, Thebaut C, Audureau E, Bernard A, Badie YL, Bohbot Y, Fard D, Nguyen LS, Monteil C, Biere L, Le Ven F, Canu M, Ribeyrolles S, Mion B, Bazire B, Fauvel C, Cautela J, Cambet T, Le Tourneau T, Donal E, Lafitte S, Magne J, Mansencal N, Coisne A; SIMULATOR investigators. Effectiveness of Simulation-Based Training on Transesophageal Echocardiography Learning: The SIMULATOR Randomized Clinical Trial. JAMA Cardiol. 2023 Mar 1;8(3):248-256. doi: 10.1001/jamacardio.2022.5016. PMID 37070491
- [Background] Damewood S, Jeanmonod D, Cadigan B. Comparison of a multimedia simulator to a human model for teaching FAST exam image interpretation and image acquisition. Acad Emerg Med. 2011 Apr;18(4):413-9. doi: 10.1111/j.1553-2712.2011.01037.x. PMID 21496145
- See also: Official page of the Advanced Medical Simulation Center at the University of Turin, providing resources and information about simulation-based medical education — https://www.dsm.unito.it/do/home.pl/View?doc=/didattica/Centro_di_simulazione_medica_avanzata.html